CLINICAL TRIAL: NCT01988896
Title: A Phase Ib Study of the Safety and Pharmacology of Atezolizumab Administered With Cobimetinib in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of Atezolizumab in Combination With Cobimetinib in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP28363; 2013-003329-27 (EudraCT Number)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-Escalation: Cobimetinib, Atezolizumab (Experimental): Participants will receive single dose of 800 milligrams (mg) of atezolizumab IV infusion on Day 1, 15 and 29 of Cycle 1 (cycle length=42 days [14-day run-in period + 28-day concomitant dosing period]), thereafter with atezolizumab IV dosing every 2 weeks (q2w) in all subsequent treatment cycles (28 days each). Combination with cobimetinib will begin on Cycle 1 Day 15 and will be given at increasing dose levels during Stage 1. During Stage 1, cobimetinib will be administered once daily (QD) orally for 21 consecutive days out of 28 days (21/7 dosing schedule) at a starting dose of 20 mg with escalation of 20 mg until the maximum tolerated dose (MTD; not more than 60 mg) for the two-drug combination.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Dose-Expansion: Cobimetinib, Atezolizumab (Experimental): Participants will receive single dose of 800 mg of atezolizumab IV infusion q2w in all subsequent treatment cycles (28 days each). Participants will receive cobimetinib at the selected recommended RP2D on Days 1-14 of each 28-day cycle during Stage 2.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered at a fixed dose as specified via IV infusion.
  Other Names: MPDL3280
Drug: Cobimetinib — Cobimetinib will be administered orally at an escalating dose during Stage 1 and at RP2D during Stage 2.
  Other Names: GDC-0973

SUMMARY:
This is a Phase Ib, open-label, multicenter study designed to assess the safety, tolerability, and pharmacokinetics of coadministration of intravenous (IV) dosing of atezolizumab (an engineered anti-programmed death-ligand 1 [anti-PD-L1] antibody) and oral dosing of cobimetinib in participants with metastatic or locally advanced cancer for which no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor that is metastatic, locally advanced or recurrent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Measurable disease, as defined by RECIST v 1.1
* Adequate hematologic and end organ function
* Use of highly effective contraception
* Histological tumor tissue specimen
* Participants enrolling in the indication-specific expansion cohorts in Stage 2 must consent to tumor biopsies and must have one of the following types of cancer:

  * Metatastic colorectal cancer
  * Non-small cell lung cancer
  * Melanoma

Exclusion Criteria:

Cancer-Specific Exclusion Criteria:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Known active or untreated central nervous system (CNS) metastases
* Leptomeningeal disease
* Uncontrolled tumor-related pain or uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent (once monthly or more frequently) drainage procedures
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab

General Medical Exclusion Criteria:

* Pregnant and lactating women
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cell or any component of the atezolizumab formulation
* History of autoimmune disease
* Participants with prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus (HIV)
* Participants with active hepatitis B, hepatitis C, or tuberculosis
* Severe infections within 4 weeks prior to Cycle 1 Day 1
* Signs or symptoms of infection within 2 weeks prior to Cycle 1 Day 1
* Received therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* Significant cardiovascular disease
* Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1 Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1

Exclusion Criteria Unique to Cobimetinib:

* History of prior significant toxicity from another mitogen-activated protein kinase (MEK) pathway inhibitor requiring discontinuation of treatment
* Allergy or hypersensitivity to components of the cobimetinib formulations
* History of congenital long QT syndrome or corrected QT interval (QTc) greater than (>) 450 milliseconds at screening
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower, as determined by echocardiogram or Multi Gated Acquisition Scan (MUGA) scan
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* History of malabsorption syndrome or other condition that would interfere with enteral absorption

Exclusion Criteria Related to Medications:

* Prior treatment with clusters of differentiation (CD) 137 agonists or immune checkpoint blockade therapies, systemic immunostimulatory agents, or systemic immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-12-27 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Phase I: Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Day 15 to Day 42 of Cycle 1 (cycle length=42 days) of dose-escalation phase
Phase I: Maximum Tolerated Dose of Cobimetinib | Day 15 to Day 42 of Cycle 1 (cycle length=42 days) of dose-escalation phase
Phase I: Recommended Phase II Dose of Cobimetinib when Combined with Atezolizumab | Day 15 to Day 42 of Cycle 1 (cycle length=42 days) of dose-escalation phase

SECONDARY OUTCOMES:
Percentage of Participants With Anti-Therapeutic Antibody (ATA) Response to Azetolizumab | Pre-infusion (Hour 0) on Day 1 of Cycles 1, 2, 3, 4, 8 (cycle length=42 days for Cycle 1; 28 days for subsequent cycles) and at treatment completion visit (up to approximately 3.5 years)
Percentage of Participants With Adverse Events (AEs) or Serious AEs (SAEs) | Baseline up to approximately 3.5 years
Serum Maximum Concentration (Cmax) of Atezolizumab | Pre-infusion (Hour 0) on Day 1 of Cycles 2, 3, 4, 8 (cycle length=28 days) and at treatment completion visit (up to approximately 3.5 years); 30 minutes post-infusion (duration=60 minutes) on Cycle 1 Day 1 (cycle length=42 days)
Serum Minimum Concentration (Cmin) of Atezolizumab | Pre-infusion (Hour 0) on Day 1 of Cycles 2, 3, 4, 8 (cycle length=28 days) and at treatment completion visit (up to approximately 3.5 years)
Plasma Cmax of Cobimetinib | Pre-dose (Hour 0) and Hours 2, 4, 6 post-dose on Day 29 of Cycle 1 (cycle length=42 days) and Day 15 of Cycle 2 (cycle length=28 days)
Plasma Cmin of Cobimetinib | Pre-dose (Hour 0) on Day 29 of Cycle 1 (cycle length=42 days) and Day 15 of Cycle 2 (cycle length=28 days)
Area Under the Concentration-Time Curve (AUC) of Cobimetinib | Pre-dose (Hour 0) and Hours 2, 4, 6 post-dose on Day 29 of Cycle 1 (cycle length=42 days) and Day 15 of Cycle 2 (cycle length=28 days)
Percentage of Participants With Best Overall Response, as Determined by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Baseline up to 3.5 years (detailed time frame is provided in the description)
  Baseline up to 3.5 years (assessed at Baseline then every 8 weeks for the first 48 weeks following Day 1 of Cycle 1 [cycle length=42 days]; thereafter every 12 weeks until progressive disease [PD] or death due to any cause, whichever occurs first [up to approximately 3.5 years])
Percentage of Participants With Objective Response (OR; Confirmed Complete Response or Partial Response) as Assessed by Investigator Using RECIST v1.1 | Baseline up to 3.5 years (assessed at Baseline then every 8 weeks for the first 48 weeks following Day 1 Cycle 1 [cycle length=42 days]; thereafter every 12 weeks until PD or death due to any cause, whichever occurs first [up to approximately 3.5 years])
Duration of OR, as Determined by Investigator Using RECIST v1.1 | Baseline up to 3.5 years (assessed at Baseline then every 8 weeks for the first 48 weeks following Day 1 Cycle 1 [cycle length=42 days]; thereafter every 12 weeks until PD or death due to any cause, whichever occurs first [up to approximately 3.5 years])
Progression-Free Survival (PFS), as Determined by Investigator Using RECIST v1.1 | Baseline up to 3.5 years (assessed at Baseline then every 8 weeks for the first 48 weeks following Day 1 Cycle 1 [cycle length=42 days]; thereafter every 12 weeks until PD or death due to any cause, whichever occurs first [up to approximately 3.5 years])
Overall Survival (OS) | Baseline up to death due to any cause (up to approximately 3.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (11):
  - Stanford University Medical Center, Palo Alto, California
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Massachusets General Hospital Clinical Trial Network and Institute, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr; Neurology/MS Center, Boston, Massachusetts
  - Sloan Kettering Cancer Center; Pediatric Hematology/Oncology, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Compass Oncology, Portland, Oregon
  - SCRI-Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, P.A., Arlington, Texas
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- Australia (2):
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (3):
  - Princess Margaret Hospital; Department of Med Oncology, Toronto, Ontario
  - CHUM Hôpital Notre-Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Germany (2):
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- National University Hospital; Cancer Center, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul

REFERENCES:
- [Derived] Hellmann MD, Kim TW, Lee CB, Goh BC, Miller WH Jr, Oh DY, Jamal R, Chee CE, Chow LQM, Gainor JF, Desai J, Solomon BJ, Das Thakur M, Pitcher B, Foster P, Hernandez G, Wongchenko MJ, Cha E, Bang YJ, Siu LL, Bendell J. Phase Ib study of atezolizumab combined with cobimetinib in patients with solid tumors. Ann Oncol. 2019 Jul 1;30(7):1134-1142. doi: 10.1093/annonc/mdz113. PMID 30918950